CLINICAL TRIAL: NCT03075020
Title: Basic Research on Carbon Monoxide's Headache Inducing Characteristics in a Humane Experimental Headache Model
Brief Title: Carbon Monoxide Migraine-inducing Effects in Patients With Migraine Without Aura.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Hashmat Ghanizada, MD, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-16021497
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Carbon Monoxide; Air

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active carbon monoxide (Active Comparator): Inhalation of carbon monoxide up to a carboxyhemoglobin concentration 22%
  Interventions: Other: Carbon monoxide
- Air (Placebo Comparator)
  Interventions: Other: AIR

INTERVENTIONS:
Other: Carbon monoxide — carbon monoxide, 4.7, Purity 99.997, inhalation of carbon monoxide in a volume corresponding to carboxyhemoglobin 10 and 20%, calculated from baseline Hg and body mass
  Arms: Active carbon monoxide
Other: AIR — Room air will be administered as placebo
  Arms: Air

SUMMARY:
To investigate headache score and accompanying symptoms during and after inhalation of carbon monoxide.

DETAILED DESCRIPTION:
To investigate headache score and accompanying symptoms during and after inhalation of carbon monoxide.

With transcranial Doppler imaging, c-scan and laser speckle the investigators will investigate changes in blood flow velocity of the middle cerebral artery (MCA), diameter of the superficial temporal artery (STA), the radial artery and facial skin perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-50
* 50-100 kg

Exclusion Criteria:

* Tension type headache more than once/month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the halflife for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Headache within the last 24 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease
* Smoking
* Primary relatives with current or previous migraine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Headache scores, 12 hours | 12 hours
  Comparison between carbon monoxide and placebo (atmospheric air)

SECONDARY OUTCOMES:
Facial blood flow | [ Time Frame: 0-180 min ]
  Carbon monoxide induced changes in facial blood flow before and after inhalation.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No